CLINICAL TRIAL: NCT06277479
Title: Late Effects and Health-Related Quality of Life in Survivors of Allogeneic Hematopoietic - a Cross-sectional Study
Brief Title: Late Effects and HRQoL in Survivors of Allo-HSCT - a Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Mette Schaufuss Engedal, Clinical nurse specialist, Ph.d student, Rigshospitalet, Denmark
Other Study IDs: Rigshospitalet. Hematology
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hematological Diseases
Keywords: Late effects. Survivorship. Allo-HSCT
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AlloHSCT Rigshospitalet: All patients treated at Department of Hematology, Rigshospitalet
- AlloHSCT Skejby: All patients treated at Department of Hematology, Skejby

SUMMARY:
The cross-sectional study aims to describe the burden of late effects and survivorship-specific health-related quality of life in a nationwide cohort of patients treated with allo-HSCT in Denmark. Further, identify demographic, medical or personal factors associated with better self-reported health and quality of life.

DETAILED DESCRIPTION:
Objective

The cross-sectional study aims to describe the burden of late effects and survivorship-specific health-related quality of life in a nationwide cohort of patients treated with allo-HSCT in Denmark. Further, identify demographic, medical or personal factors associated with better self-reported health and quality of life.

Method

An observational, descriptive, cross-sectional study using clinical data and self-reported questionnaires to assess the occurrence of comorbidities and self-reported late effects in survivors treated with allo-HSCT in Denmark between 1970 and 2024.

Study population

All survivors treated for malignant or non-malignant hematological disease with allo-HCST at the age of 18-79 years from 1970-2024 in Denmark are eligible (n=1.436).

Endpoints

* Self-reported survivorship specific HRQoL measured by EORTC-QOL- Survivorship 100.
* Degree of health literacy measured by the Health Literacy Questionnaire (HLQ).
* Occurrence or degree of Chronic Graft Versus Host Disease measured by modified Lee Chronic Graft versus host disease Symptom Scale.

ELIGIBILITY:
Inclusion Criteria:

* All survivors treated for malignant or non-malignant hematological disease with allogeneic hematopoietic stem cell transplantation at the age of 18-79 years from 1970-2024 in Denmark are eligible

Exclusion Criteria:

* Patient unable to read and understand danish are excluded from study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All survivors treated for malignant or non-malignant hematological disease with allogeneic hematopoietic stem cell transplantation at the age of 18-79 years from 1970-2024 in Denmark are eligible
Sampling Method: Non-Probability Sample
Enrollment: 1262 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
EORTC Quality of Life Survivorship Core questionnaire (EORTC-QOL-SURV100) | may 2024 - August 2024
  The QLQ-SURV100 is based on the EORTC Quality of Life core questionnaire (QLQ-C30). Applicable to disease-free cancer survivors. It consists of 100 questions divided over thirteen functional scales (i.e. Physical; Role ; Emotional; and Cognitive functioning; Body image; Symptom awareness; Positive health behavior change; Positive life outlook; Positive impact on behavior towards others; Positive social functioning; Work; Sexual functioning; Global health status), nine symptom scales (i.e. Social isolation; Fatigue; Pain; Sleep problems; Health distress; Negative health outlook; Social interference; Sexual problems), one Symptom checklist assessing chronic side effects of cancer treatments, and twelve single items.
  Score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QL represents a high QL, but a high score for a symptom item represents a high level of symptomatology.

SECONDARY OUTCOMES:
Health literacy Questionnaire (HLQ) | may 2024 - august 2024
  The HLQ consists of 9 scales representing 9 dimensions of health literacy. Each HLQ scale has 4-6 items. The HLQ does not provide one overall summative score. The 9 scale scores will reflect a person's strengths and needs in the different dimensions of health literacy.Higher score reflect a higher degree of health literacy.
  1. Feeling understood and supported by healthcare providers
  2. Having sufficient information to manage my health
  3. Actively managing my health
  4. Social support for health
  5. Appraisal of health information
  6. Ability to actively engage with healthcare providers
  7. Navigating the healthcare system
  8. Ability to find good health information
  9. Understand health information well enough to know what to do.
Modified 7-day Lee Chronic-versus-Host Disease Symptom Scale | may 2024 - august 2024
  The Modified 7-day Lee Chronic-versus-Host Disease Symptom Scale is a validated questionnaire to measure degree of Graft Versus Host disease. The scale contains 28 items grouped in 7 subscales (skin, eye, mouth, lung, nutrition, energy, and psychological). Patients report how "bothered" they feel about each symptom over the previous 7 days using a five-point Likert scale from "not at all" to "extremely". Score range from 0 to 100, with a higher score indicating worse symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mette Schaufuss Engedal, MSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Mette Schaufuss Engedal, Copenhagen, Denmark